CLINICAL TRIAL: NCT02545673
Title: Enhanced Linkage to HIV Care Following Home-Based HIV Testing in Rural Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susan M Kiene (Other)
Collaborators: Makerere University (Other); University of Connecticut (Other); Harvard School of Public Health (HSPH) (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Susan M Kiene, Professor, San Diego State University
Organization: San Diego State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UG2015_01; R01MH106391 (NIH)
Record Dates: First submitted 2015-08-31; First posted 2015-09-10 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: HIV
Keywords: Intervention Studies; Access to Health Care; Social Stigma; Social Support
MeSH Terms: conditions — Social Stigma | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Linkage (Experimental): Participants will receive the enhanced linkage to care Intervention. Behavioral: Enhanced linkage to care Intervention Multiple sessions will focus on providing orientation to the HIV care system, counseling to help clients identify and reduce barriers to engagement in care, assistance disclosing and identifying a treatment supporter, and stigma reduction through increasing social support. The approach is guided by the HIV Stigma Framework.
  Interventions: Behavioral: Enhanced linkage to care
- Standard-of-care plus (Active Comparator): Behavioral: Participants will receive the standard-of-care (paper-based referrals) plus return of CD4 test results to their home.
  Interventions: Behavioral: Standard-of-care plus

INTERVENTIONS:
Behavioral: Enhanced linkage to care
  Arms: Enhanced Linkage
Behavioral: Standard-of-care plus
  Arms: Standard-of-care plus

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a linkage to care intervention at achieving HIV viral suppression and intermediate outcomes of linkage/time to care, time to /receipt of opportunistic infection prophylaxis, and antiretroviral therapy (ART) among people testing HIV positive during home-based HIV counseling and testing (HBHCT) in rural Uganda.

DETAILED DESCRIPTION:
Throughout sub-Saharan Africa there is a pressing need to facilitate early and easier entry into HIV care and treatment; up to two-thirds of patients are lost to follow up between testing HIV positive and initiation of antiretroviral (ARV) treatment. Home-based HIV testing and counseling (HBHCT), which identifies those who are HIV positive at earlier disease stages than other testing approaches, is becoming a large component of many sub-Saharan African countries' HIV prevention programs, including Uganda's. Paper-based referral to care, sometimes adding follow-up home visits, is the most common linkage-to-care approach with HBHCT. Linkage to care may be challenging with HBHCT since the testing occurs in the home at a distance from a health facility. The investigators propose to test an intervention which enhances a linkage to care intervention tested in an urban Ugandan provider-initiated HIV testing setting and found to improve linkage to care. The aims of the project are: (1) In a cluster randomized trial compare the effectiveness of the enhanced linkage to care intervention vs. standard-of-care (paper based referrals) at achieving HIV viral suppression and intermediate outcomes of linkage to care, receipt of opportunistic infection prophylaxis, and ART initiation among those eligible for antiretroviral therapy (ART). (2) Using the standard-of-care group as a natural history control, collect longitudinal data on barriers to and facilitators of linkage to and retention in care and treatment and HIV viral suppression. (3) Estimate the cost-effectiveness of the intervention, as compared to standard-of-care, in terms of major study outcomes.

Participation in the full study will last 12 months. All participants will first undergo HBHCT, viral load and CD4 testing, and complete a brief questionnaire. Participants will then be randomly assigned to one of two study arms: the enhanced linkage to care intervention arm or the standard-of-care control arm. Participants in both study arms will participate in interviewer administered questionnaires at 6 months and 12 months follow-up, viral load and CD4 testing at 12 month follow-up, and will permit the research team to access their medical records to extract information about their health status and linkage to care. Participants in the intervention arm will also receive a series of counseling sessions with an HIV counselor taking place at the participant's home, clinic, and over the phone. These sessions will last approximately 30 minutes, and consist of counseling to help clients identify and reduce barriers to engagement in care, assistance disclosing and identifying a treatment supporter, and stigma reduction through increasing social support.

ELIGIBILITY:
Inclusion/Exclusion for home-based HIV counseling and testing and brief baseline questionnaire:

Inclusion Criteria:

• 18-59 years of age or an emancipated minor

Exclusion Criteria:

* not a resident of the household
* Does not speak Luganda or English

Inclusion/Exclusion for the Intervention Study:

Inclusion criteria:

* participated in the baseline interview and home-based HIV counseling and testing,
* newly diagnosed HIV positive in the home-based HIV counseling and testing or previously diagnosed but never linked to HIV care

Exclusion criteria:

• Other household members also newly diagnosed as HIV positive/previously diagnosed but never linked to care. Only one person per household will be eligible to enroll

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 567 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Undetectable HIV Viral load | 12 months follow up
  defined as HIV RNA <20 cells/ml collected via venous blood draw

SECONDARY OUTCOMES:
HIV Viral load Suppression | 12 months follow up
  defined as HIV RNA <1000 cells/ml collected via venous blood draw
Linkage to HIV care | 6 and 12 months follow up
  Enrollment in an HIV clinic with a 2nd clinic visit
Initiating ART | 6 and 12 months follow up
  Percentage of eligible participants initiating ART
Short-term retention on treatment | 6 and 12 months follow up
  on ART at 6 and 12 month follow up: reporting taking ART at each follow-up
Time to HIV care | 6 and 12 months follow up
  Time from HIV testing to enrollment in an HIV clinic
Time to receipt of ART | 6 and 12 months follow up
  Time from HIV testing to receipt of ART
Short-term retention in care: Missed visits | 6 and 12 months follow up
  Missed visit count: number of missed visits accrued (count measure) based on scheduled visits determined by Ministry of Health clinical guidelines
Short-term retention in care: Proportion of kept visits/scheduled visits | 6 and 12 months follow up
  Proportion of kept visits/scheduled visits (kept + missed visits)
Short-term retention in care: 4 month visit constancy | 6 and 12 months follow up
  4-month constancy 4 month visit constancy: number of 4-month intervals with at least 1 kept visit

OTHER OUTCOMES:
Receipt of co-trimoxazole | 6 and 12 months follow up
  The percentage of participants who received co-trimoxazole
Time to receipt of co-trimozazole | 6 and 12 months follow up
  Time to receipt of co-trimoxazole

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Kiene, PhD, Principal Investigator — San Diego State University
Locations (1):
- Butambala, Mpigi, Mityana, Gomba Districts, Gombe, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with researchers within study investigators' institutions and with other researchers upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Data will be available to other researchers 2 years after publication of the trial results.
Access Criteria: Contact principal investigators Drs. Kiene or Wanyenze to request access.

REFERENCES:
- [Derived] Kiene SM, Kalichman SC, Sileo KM, Menzies NA, Naigino R, Lin CD, Bateganya MH, Lule H, Wanyenze RK. Efficacy of an enhanced linkage to HIV care intervention at improving linkage to HIV care and achieving viral suppression following home-based HIV testing in rural Uganda: study protocol for the Ekkubo/PATH cluster randomized controlled trial. BMC Infect Dis. 2017 Jul 3;17(1):460. doi: 10.1186/s12879-017-2537-z. PMID 28673251